CLINICAL TRIAL: NCT04284657
Title: Pravastatin and Alkali Therapy in Patients With Autosomal Dominant Polycystic Kidney Disease
Acronym: ADPKD-SAT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Nuria M. Pastor-Soler, Associate Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-18-00170
Record Dates: First submitted 2019-04-11; First posted 2020-02-26 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease
Keywords: Polycystic Kidney Disease; ADPKD; PKD
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Polycystic Kidney Diseases | interventions — Pravastatin; Sodium Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- ARM I: Control group (No Intervention): Standard therapy alone
- ARM II: PRAVASTATIN (Active Comparator): Standard therapy and PRAVASTATIN 40 mg QD
  Interventions: Drug: Pravastatin
- ARM III: PRAV + Sodium Citrate (Active Comparator): Standard therapy and PRAVASTATIN 40 mg QD and Sodium Citrate (up to 30 mL TID)
  Interventions: Drug: Pravastatin; Drug: sodium citrate

INTERVENTIONS:
Drug: Pravastatin — Pravastatin 40 mg QD
  Arms: ARM II: PRAVASTATIN; ARM III: PRAV + Sodium Citrate
Drug: sodium citrate — sodium citrate up to 30 ml TID
  Arms: ARM III: PRAV + Sodium Citrate

SUMMARY:
This is an one-year open-label study to determine treatment efficacy and feasibility of a trial that uses open-label interventions in ADPKD patients.

DETAILED DESCRIPTION:
Polycystic Kidney Disease (PKD) is the most common genetic disease leading to End Stage Kidney Disease (ESKD), affecting between 1 in 500-1000 individuals from every ethnic group. The autosomal dominant (ADPKD) form arises from a two-hit downregulation of proteins encoded by either PKD1 or PKD2. Although many potential therapies have been studied to slow progression of ADPKD, none to date have been proven to be both safe and effective in slowing disease progression. Cholesterol-lowering agents called statins have shown promise in the treatment of younger ADPKD patients, reducing inflammation and progression as assessed by kidney growth, but their utility appears to be limited in older populations and those with more advanced chronic kidney disease (CKD). Recent evidence suggests that acidosis, as often seen in patients with worsening CKD and which may enhance CKD progression, limits the effectiveness of statins and enhances their potential toxicity. The investigators thus hypothesize that correction of acidosis along with statin treatment will be a safe and effective therapeutic regimen to slow CKD progression in the adult ADPKD population and improve overall quality of life in these patients. To test this hypothesis, the investigators will conduct a pilot open-label randomized clinical trial in ADPKD patients with estimated GFR >45 min (Stage 1-3a CKD) comparing three treatment groups: control, pravastatin (40 mg po qd), and pravastatin plus sodium citrate solution (30 mL po total daily dose) over one year. During the study period, through study visits along with serial blood draws and urinary measurements, the investigators will evaluate safety and tolerability of these treatment regimens, follow renal function and investigate the role of these treatments on acidosis, inflammatory and metabolic biomarkers in patients enrolled at an outpatient facility. This study will establish the framework for larger clinical trials in ADPKD. Moreover, if the results of this study suggest safety/tolerability or potential benefits of statins and alkali therapy in this ADPKD population, the investigators will seek extramural funding for a larger clinical trial to test this therapeutic strategy in ADPKD.

ELIGIBILITY:
Inclusion Criteria:

1. Patient voluntarily gives informed consent to participate in the study and signed study's IC and HIPAA.
2. Patient is age 18 or older at the time of consent.
3. If applicable, female of reproductive potential (Females who are successfully sterilized (surgical sterilization methods include hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or are postmenopausal (defined as amenorrhea for at least 12 consecutive months) are not considered to be of reproductive potential) must be non-pregnant (as confirmed by a urine pregnancy test at screening) and non-lactating, and agree:

   1. Either abstain from intercourse (when it is in line with their preferred and usual lifestyle), or
   2. Use 2 medically acceptable, highly-effective forms of contraception for the duration of study, and at least 30 days after discontinuing study drug (highly-effective forms of contraception can include approved hormonal contraceptives (oral, injectable, and implantable), and barrier methods (such as a condom or diaphragm) when used with a spermicide.))
4. Patients has ADPKD diagnosed by unified criteria using a combination of ultrasound results, genotyping and MRI as needed (1, 2). Kidney ultrasound is usually used for screening because it is safe, effective, and inexpensive. Diagnostic criteria are based upon whether the genotype is known. Disease severity varies between the different genotypes. The great majority of patients at risk for ADPKD are from families with an unknown genotype. This diagnosis will take place prior to recruitment / inclusion into the study.

   The following ultrasonographic criteria for the diagnosis of ADPKD are for at-risk patients from families of where the genotype is not known:
   1. If the patient is between 18 and 39 years of age, at least three unilateral or bilateral kidney cysts. The specificity and positive predictive value at this age-range is 100 percent. (sensitivity of 82 and 96 percent for individuals between 15 and 29 years and between 30 to 39 years of age, respectively).
   2. If the patient is 40 to 59 years of age, at least two cysts in each kidney (sensitivity, specificity, and positive predictive value of 90, 100, and 100 percent, respectively).
   3. Among individuals 60 years or older, at least four cysts in each kidney. (100 percent sensitivity and specificity).
5. The above patients with estimated GFR ≥30 ml/min i.e. with stage 1-3b CKD
6. Plasma bicarbonate ≤ 25 mMol/L
7. Metabolic acidosis
8. The patient agrees to immediately inform Investigator and research coordinator of any changes or planned changes in concomitant medication

Exclusion Criteria

1. Patients with known allergy or sensitive to Pravastatin or NaCitrate
2. Acute coronary disease, liver disease, muscle disease, or a history of pulmonary edema
3. Creatine Phospho Kinase (CPK) > 2ULN (2.5 ULN in African Americans). Elevated creatine phosphokinase could be a marker of rhabdomyolysis, which is a potential side effect of pravastatin. In general, patients with African American ancestry can have higher normal level of CPK
4. Patients with systemic disease that impacting kidney per Investigator's decision
5. Patients with known unstable cerebral aneurysm per Investigator's decision
6. Pregnancy or lactation, or patients who refuse to use recommended contraception methods
7. Proteinuria > 500 mg/day
8. History of non-compliance of medication per Investigator's decision
9. Patients with uncontrolled hypertension, edema, or development of severe MA as per Investigator's decision
10. History of cancer
11. History of liver disease: hepatic failure/shock, cirrhosis
12. Current or planned use of any of prohibited concomitant medication
13. Patients with history of nephrolithiasis

Following medications prohibited at the time of enrollment and during the study and if the patient is started on these medications then the patient will be excluded from the study:

* rapamycin or its analogues
* tolvaptan
* spironolactone
* cimetidine and ketoconazole
* erythromycin
* cyclosporine
* gemfibrozil
* colchicine
* niacin (>1 g/day)
* other lipid lowering medications in the class of statins

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2025-08-04 (Actual); Study Completion 2025-08-04 (Actual)

PRIMARY OUTCOMES:
Changes in kidney function in patients enrolled in different arms of the study | 12 months
  The investigators will estimate the effect of Pravastatin and NaCitrate on kidney function in patients with ADPKD compared to Pravastatin alone or Standard therapy: serum creatinine and serum blood urea nitrogen, serum electrolytes contribute to evaluate kidney function.
Changes in liver function in patients enrolled in different arms of the study | 12 months
  The investigators will test liver function test panels in patients with ADPKD compared to Pravastatin alone or Standard therapy. The liver function panel should be within normal limits for enrollment and continuation in the study. Liver function tests include AST > 3ULN, ALT > 3ULN, Total Bilirubin > 2 ULN, or increase in prothrombin time to abnormal level INR >1.5 repeated two weeks apart
Changes in blood pressure in patients enrolled in different arms of the study | 12 months
  The investigators will estimate the effect of Pravastatin and NaCitrate on blood pressure (systolic and diastolic) in patients with ADPKD compared to Pravastatin alone or Standard therapy
Changes in muscle injury marker function in patients enrolled in different arms of the study | 12 months
  The investigators will estimate the effect of Pravastatin and NaCitrate on creatine phospho kinase (CPK) in patients with ADPKD compared to Pravastatin alone or Standard therapy.
Changes in muscle tenderness in patients enrolled in the study | 12 months
  The investigators will estimate the effect of Pravastatin and NaCitrate on muscle tenderness in patients with ADPKD compared to Pravastatin alone or Standard therapy. The physical exam will evaluate tenderness to palpation in major muscle groups such as leg, arm and back muscles. It will be graded as presence or absence. The patients will only be enrolled if there is absence of tenderness in muscles upon palpation on physical exam. If there is tenderness on exam or the patient reports tenderness that is then confirmed by exam the patient will be removed from the study.

SECONDARY OUTCOMES:
Urinary alkalinization changes | 12 months
  These parameters will be ascertained by measurements of urinary pH and serum electrolytes.
Inflammatory markers in blood and urine | 12 months
  The investigators will assess inflammatory markers (interleukins, prostaglandins and other cytokines) in leukocytes, plasma, and urine in the different study groups.
  The biomarkers that will be measured are
  HETE / HODE species phospho-AMPK Inflammatory and metabolic biomarkers: NGAL, KIM1 in blood and urine
AMPK pathway activation | 12 months
  The investigators will determine whether and to what extent the AMPK pathway is activated in leukocytes and urine derived from patients in the study groups at the different study visits, and correlate AMPK activation with biological effects.

CONTACTS AND LOCATIONS:
Locations (1):
- Keck School of Medicine of University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No